CLINICAL TRIAL: NCT06016491
Title: The Effect of Acupressure on Menopausal Symptoms: A Randomized, Sham Controlled Study
Brief Title: The Effect of Acupressure on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Melek Yesil Bayulgen, Lecturer (Principal Investigator), Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin Univers
Record Dates: First submitted 2023-08-16; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Menopause; Acupressure
Keywords: Menopause; Acupressure; Menopausal symptoms
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: 81 people who attended the menopause school and met the inclusion criteria were selected by simple random sampling. Each of the women was allowed to draw from the numbers in the bell, and those who drew odd numbers were assigned to the placebo group, and those who drew even numbers were assigned to the acupressure group. Acupressure pressure point was applied to all women included in the study. Participants were blinded because they did not know whether the women were given acupressure or placebo acupressure. Researchers could not be blinded because they were also practitioners (Melek Yeşil Bayülgen and Fatma Hikmet Yeşil). When the research was completed, the data were analyzed by a statistician who did not know the groups and the findings were reported
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): Before the acupressure application, the woman to be applied was informed in a quiet room for ease of application, and then she was ensured to be in a comfortable position. Women were taught to practice on a total of two points, the kidney meridian (Yong Quan-KD1) and the spleen meridian (Sanyinjiao-SP6). Since the symmetry of the selected two different points on the other extremity will also be applied, a total of 8 minutes of compression was applied to each point, provided that it was two minutes. Depending on the preparation and compression time on each point, an average of 10 minutes was applied to each patient, and then the patients were asked to apply it to themselves. After making sure that the women learned, they were asked to apply acupressure on their own. They applied a total of 12 sessions, three times a week for a total of four weeks. To remind the session day, information was given by the researcher via short message.
  Interventions: Behavioral: acupressure
- Sham acupressure group (Sham Comparator): After all the preparations (suitability of sound and environment and information) before the application to the acupressure group were made in the sham group, the sham acupressure points determined parallel to the KD1 and SP6 points (approximately 1-1.5 cm away) were put on the bone area where the meridians do not pass has been applied.
  Similar to the acupressure group, the sham acupresuure group was treated with symmetrical extremities and for similar durations.
  Interventions: Behavioral: Sham acupressure

INTERVENTIONS:
Behavioral: acupressure — Depending on the preparation and compression time on each point, an average of 10 minutes was applied to each woman, and then the person were asked to apply it to themselves. After making sure that the women learned, they were asked to apply acupressure on their own. They applied a total of 12 sessions, three times a week for a total of four weeks.
  Arms: Acupressure group
Behavioral: Sham acupressure — Compression was applied on the bone region where the meridians did not pass, parallel to the KD1 and SP6 points (approximately 1-1.5 cm away). Similar to the acupressure group, the sham group was treated with symmetrical extremities and for similar durati
  Arms: Sham acupressure group

SUMMARY:
This is a prospective, randomized, placebo-controlled and single-blind study planned to determine the effect of acupressure application on menopausal symptoms.

The hypothesis of the study is that acupressure reduces women's menopausal symptoms.

DETAILED DESCRIPTION:
Menopause is a physiological process during which most women have difficulties and face many problems. Acupressure can be taught and used safely as an effective method to manage the symptoms that women experience during menopause.

This study aims to determine the effect of acupressure on menopausal symptoms. The study has a prospective, randomized, sham-controlled, single-blind design. The research was conducted with 81 women (acupressure n=40, sham acupressure n=41) attending the "Menopause School" in a public hospital in Türkiye between July 05, 2021 and August 02, 2021. Both groups received acupressure application thrice a week for four weeks, 12 sessions in total. The data was obtained using a personal information form and a Menopause Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish
* No psychiatric illness
* Natural menopause
* Not on hormone replacement therapy
* Women who volunteered to participate in the study and did not receive any integrated therapy were included.

Exclusion Criteria:

* Those who have undergone menopause with the surgical method
* For lower extremity vascular disease, fracture, sprain or injury, diabetes, cardiovascular disease, thyroid disease, etc. with a diagnosis
* Women who received any integrative therapy were not included in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | Change from before implementation, 0th week and 4th week of practice
  Menopause symptom rating scale was used to evaluate menopausal symptoms. The Turkish reliability and validity study was conducted by Can (2005). The scale consists of 11 items and 3 sub-dimensions. For each item, there are "0=None", "1=Mild", "2=Moderate", "3=Severe" and "4=Very Severe" options. Sub-dimensions of the scale; somatic complaints (items 1,2,3 and 11), psychological complaints (items 4,5,6 and 7), and urogenital complaints (items 8,9 and 10). The total score of the scale ranges from 0 to 44. The somatic complaints sub-dimension is scored between 0-16, the psychological complaints sub-dimension 0-16, and the urogenital complaints sub-dimension 0-12. An increase in the total score obtained from the scale indicates that the severity of the complaints increases and the quality of life is negatively affected.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No